CLINICAL TRIAL: NCT02731053
Title: Pilot Effectiveness Trial of the French Blues Indicated Depression Prevention Program
Brief Title: Effectiveness Trial of the French Blues Indicated Depression Prevention Program
Acronym: French Blues
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Université de Montréal (Other)
Responsible Party: Principal Investigator, Frédéric N. Brière, PhD, Principal Investigator, Université de Montréal
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: FRQSC2016-NP-191870
Record Dates: First submitted 2016-03-15; First posted 2016-04-07 (Estimated); Last update posted 2017-09-28 (Actual); Status verified 2017-09

CONDITIONS: Depression
Keywords: Depression; Prevention; Adolescents; School; Effectiveness
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Blues program (Experimental): Participants will attend 6 weekly 1-hour sessions of group cognitive-behavioral therapy administered by school staff, and will do home practice between sessions and after the program individually using a web site (called the Blues App)
  Interventions: Behavioral: Blues program
- Control (No Intervention): Participants will receive a brochure describing the nature, causes, and consequences of depression, as well as available prevention/treatment options

INTERVENTIONS:
Behavioral: Blues program — Participants will attend 6 weekly 1-hour sessions of group cognitive-behavioral therapy administered by school staff, and will do home practice between sessions and after the program individually using a web site (called the Blues App)
  Arms: Blues program

SUMMARY:
The purpose of this pilot study is to test the effectiveness of French adaptation of the Blues program, a school-based indicated depression prevention intervention. The program will be delivered by the endogenous psycho-social staff of 3 Montreal secondary schools to adolescents with sub-clinical depressive symptoms and compared to a no-intervention (Informational Brochure only) control condition, designed to represent the "usual intervention" in these schools.

ELIGIBILITY:
Inclusion Criteria:

* Elevated depressive symptoms (score of 20 or above on the Center for Epidemiological Studies - Depression screening questionnaire)

Exclusion Criteria:

* Current major depression diagnosis
* Current active suicidal behaviors
* Being in a special school curriculum for academic or behavioral problems

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 72 (Actual)
Dates: Start 2016-03; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Number of participants who develop a major depressive episode as measured using the SCID diagnostic interview (posttest, 6 month follow-up) | 6 months
Change in depressive symptoms as measured using continuous SCID scores (baseline, posttest, 6-month follow-up) | 6 months
Change in depressive symptoms as measured using the CES-D questionnaire (baseline, posttest, 6-month follow-up) | 6 months
Change in depressive symptoms as measured using the PHQ-9 questionnaire (baseline, posttest, 6-month follow-up) | 6 months

SECONDARY OUTCOMES:
Change in social adjustment as measured using "Évaluation sociale de Soi chez les jeunes adultes" questionnaire (Michaud et al., 2006) (baseline, posttest, 6-month follow-up) | 6 months
Change in anxiety symptoms as measured using the SCAS questionnaire (baseline, posttest, 6-month follow-up) | 6 months
Change in parent-child relationship as measured using a scale from the MASPAQ questionnaire (Leblanc, 1996) (baseline, posttest, 6-month follow-up) | 6 months
Change in affective school engagement as measured using a subscale of the school engagement questionnaire (Archambault et al., 2009) (baseline, posttest, 6-month follow-up) | 6 months
Change in substance use as measured using a scale from the MASPAQ questionnaire (Leblanc, 1996) (baseline, posttest, 6-month follow-up) | 6 months
Change in delinquent behaviors as measured using a scale from the MASPAQ questionnaire (Leblanc, 1996) (baseline, posttest, 6-month follow-up) | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Frederic N Briere, PhD, Principal Investigator — Université de Montréal
Locations (1):
- Université de Montréal, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No